CLINICAL TRIAL: NCT07318545
Title: Intervention for Chronic Insufficient Sleep in Young Adult Cancer Patients and Survivors: Randomized Controlled Trial
Brief Title: Intervention for Chronic Insufficient Sleep in Young Adult Cancer Patients and Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00009801; 2R44CA254637-02 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Young adult; Cancer survivor
MeSH Terms: conditions — Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice-activated virtual assistant-delivered cognitive behavioral therapy for insomnia (Experimental): More Sleep Hours Electronic Education Program (More SHEEP) is a home-based, technology-enabled intervention that delivers cognitive behavioral therapy for insomnia (CBT-I) to young adult cancer survivors. The intervention uses a screen-free, voice-activated smart speaker integrated with adaptive smart lighting and internet use monitoring to provide CBT-I components including sleep education, sleep scheduling, behavioral recommendations, and daily sleep diary collection over a 6-week period.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Voice-activated virtual assistant-delivered sleep management skills (not CBT-I) (Active Comparator): The active comparator arm will include the same hardware as the More SHEEP system, a screen-free, voice-activated smart speaker integrated with adaptive smart lighting and internet use monitoring, but will not deliver CBT-I, it will only include skills education to improve sleep.
  Interventions: Behavioral: Sleep education and skills

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I) is a structured, evidence-based treatment that helps people change thoughts and behaviors that interfere with sleep, using techniques like stimulus control, sleep restriction, cognitive restructuring, and relaxation training.
  Arms: Voice-activated virtual assistant-delivered cognitive behavioral therapy for insomnia
Behavioral: Sleep education and skills — Daily education about building better sleep habits, sleep hygiene, diet and exercise related to sleep
  Arms: Voice-activated virtual assistant-delivered sleep management skills (not CBT-I)

SUMMARY:
Young adult cancer survivors (YACS) commonly experience chronic insomnia due to many factors such as cancer related symptoms, effects of anti-cancer therapies, co-morbid mood disorders, and/or other psychosocial and economic stressors. Cognitive behavioral therapy for insomnia (CBT-I) is the gold standard for insomnia management but remains challenging to deliver to patients due to limited numbers of trained therapists, inconvenient scheduling availability, or prohibitive therapy costs. To address this critical gap in young adult cancer survivorship, the investigators propose to develop and test efficacy of the More Sleep Hours Electronic Education Program (More SHEEP), a novel system of smart speaker, smart lighting, and specialized Wi-Fi router that delivers AI-driven CBT-I to patients at home.

DETAILED DESCRIPTION:
Insomnia - defined as difficulty falling asleep, staying asleep, or nonrestorative sleep - is often accompanied by symptoms that impair daily function such as fatigue, difficulty concentrating, and mood disturbance. Affecting up to 75% of the estimated 650,000 young adult cancer survivors in the United States, insomnia has a myriad of psychological and medical sequelae that compound late in long-term effects of cancer diagnosis and treatment, including increased risk of mortality. Cognitive behavioral therapy for insomnia (CBT-I) remains the gold standard for managing chronic insomnia. Nevertheless, widespread access to trained CBT-I providers, even in accredited sleep centers, remains elusive: trained CBT-I therapists remain limited in number and traditional in-person CBT-I therapy can be time and cost prohibitive for patients. Newer attempts to develop automated web-based CBT-I are more didactic than interactive and can involve counterproductive use of smartphone screens at bedtime that can be activating and suppress the melatonin needed for sleep. To address this critical gap in young adult cancer survivorship care, the investigators propose the More Sleep Hours Electronic Education Program (More SHEEP): a CBT-I solution using a screen-free, conversational, AI-driven smart speaker, custom lighting to plan, remind and support YACS about the changes required to overcome insomnia, and a smart router to report on bedtime screen use. They propose a multi-phase project involving active patient stakeholder input and an iterative design process that will achieve the following Specific Aims: Aim 1) maximize feasibility, usability, and acceptability of the interactive CBT-I prototype; Aim 2) finalize the prototype and conduct pilot field testing of the intervention for usability; Aim 3) conduct a randomized controlled trial to determine the impact of these integrated CBT-I components on insomnia symptoms among young adult cancer survivors compared to an attention control. Successful completion of these Aims will further their long-term goal of providing novel, affordable, available, scalable, evidence-driven solutions for moderate-severe chronic insomnia among young adult cancer survivors. Furthermore, this technology can eventually be translated to other patient populations living with cancer or other serious illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-42 at time of enrollment
* history of cancer diagnosis (any type) diagnosed at/after age 15, received all treatment before age 40
* at least 6 months from date of cancer diagnosis
* history of chronic sleep disorder with Insomnia Severity Index >/= 8

Exclusion Criteria:

* Refusal to try the study intervention
* diagnosed untreated obstructive sleep apnea syndrome, or restless leg syndrome
* narcolepsy, schizophrenia, bi-polar disorder, and/or poorly controlled psychiatric diagnoses
* disease-related prognosis of less than 6 months or currently enrolled in hospice care
* planned travel out of the continental United States during the study period.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline (Day 0) and Post Intervention (6 Weeks)
  The Insomnia Severity Index (ISI) is a validated 7-item self-reported questionnaire assessing the severity of insomnia symptoms and related daytime impairment over the past two weeks. Items are scored on a 0-4 scale, producing a total score from 0 to 28, with higher scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - General | Baseline (Day 0) and Post Intervention (6 Weeks)
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a validated self-reported questionnaire assessing health-related quality of life in patients with cancer. The 27-item instrument evaluates physical, social/family, emotional, and functional well-being, with higher scores indicating better quality of life.
Functional Assessment of Cancer Therapy - Cognitive Function | Baseline (Day 0) and Post Intervention (6 Weeks)
  The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) is a validated self-reported questionnaire assessing perceived cognitive function and cognitive-related quality of life in patients with cancer. The instrument evaluates domains including perceived cognitive impairments, perceived cognitive abilities, impact on quality of life, and comments from others, with higher scores indicating better perceived cognitive function.
Satisfaction with Assigned Study Intervention (Client Satisfaction Questionnaire) | Post Intervention (6 Weeks)
  The Client Satisfaction Questionnaire (CSQ) is a 10-item validated self-reported questionnaire assessing participant satisfaction with services received. The instrument evaluates perceived quality, usefulness, and overall satisfaction with care, with higher scores indicating greater satisfaction.
Recommendation of Assigned Intervention to Family/Friends | Post Intervention (6 Weeks)
  Likert scale of participant's self-report of how likely they are to recommend the assigned intervention to family/friends (1=not at all likely, 5=very likely)
System Usability Scale | Post Intervention (6 Weeks)
  The System Usability Scale (SUS) is a validated self-reported questionnaire assessing perceived usability of a system or technology. The 10-item instrument yields a score from 0 to 100, with higher scores indicating greater perceived usability.

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Groninger, MD, Principal Investigator — Medstar Health Research Institute

IPD SHARING:
Plan to Share IPD: Undecided